CLINICAL TRIAL: NCT02172300
Title: Effect of Tiotropium on Exercise Tolerance and Static and Dynamic Lung Volumes in COPD Patients (A Randomized Double-Blind, Placebo Controlled, Parallel Group Study)
Brief Title: Effect of Tiotropium on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.131
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tiotropium (Experimental): Tiotropium inhalation capsules via HandiHaler
  Interventions: Drug: Tiotropium inhalation capsules
- Placebo (Placebo Comparator): Placebo inhalation capsules via HandiHaler
  Interventions: Drug: Placebo inhalation capsules

INTERVENTIONS:
Drug: Tiotropium inhalation capsules
  Arms: Tiotropium
Drug: Placebo inhalation capsules
  Arms: Placebo

SUMMARY:
Study to investigate whether tiotropium therapy can increase duration of steady-state exercise by decreasing dynamic and static lung hyperinflation in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients had to have a diagnosis of COPD. Patients had to meet the following spirometric and static lung volume criteria:

  * Patients had to have relatively stable, mild (stage I according to the criteria of the American Thoracic Society (ATS); original trial protocol: moderate) to severe airway obstruction with an FEV1 less than or equal to 65% of predicted values. All patients had to have presence of lung hyperinflation as demonstrated by thoracic gas volume (TGV) / functional residual capacity (FRC) greater than or equal to 120% of predicted value as determined by body plethysmography at Visit 1 (day -15).
* Male or female patients ≥ 40 but ≤ 70 years old.
* Patients had to have a cigarette smoking history of more than 10 pack-years. A pack-year was defined as the equivalent of smoking one pack of cigarettes per day for a year.
* Patients had to be able to perform all specified procedures and maintain records during the study period as required in the protocol.
* Patients had to be able to inhale medication from the HandiHaler®.
* All patients had to sign an Informed Consent Form in accordance with Good Clinical Practice (GCP) and local legislative requirements prior to participation in the trial . i.e., prior to pre-study washout of their usual pulmonary medications.

Exclusion Criteria:

* Patients with significant diseases other than COPD were to be excluded. A significant disease was defined either as a disease, which in the opinion of the investigator might have put the patient at risk because of participation in the study or a disease, which might have influenced the results of the study or the patient's ability to participate in the study.
* Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defined a disease listed as an exclusion criterion, the patient was to be excluded.
* All patients with a serum glutamic oxaloacetic transaminase (SGOT or AST) ≥ 1.5 of the upper limit of normal range (x ULN), serum glutamic pyruvic transaminase (SGPT or ALT) ≥ 1.5 x ULN, bilirubin ≥ 1.5 x ULN, or creatinine ≥ 1.5 x ULN were excluded regardless of the clinical condition. Repeat laboratory evaluation was not to be conducted in these subjects.
* Patients with a recent history (i.e., 1 year or less) of myocardial infarction.
* Patients with a recent history (i.e., 3 years or less) of heart failure, pulmonary edema, or patients with cardiac arrhythmia (with or without symptoms) or any contraindication to exercise as indicated in Protocol Appendix four (see Section 9.5.1 and Appendices 16.1.1.1 and 16.1.1.2).
* Patients with regular use of daytime oxygen therapy. (In centers with significantly decreased barometric pressure, exercise tests can be done with inhaled oxygen).
* Patients with known active tuberculosis.
* Patients with a history of cancer within the last 5 years. Patients with treated basal cell carcinoma were allowed.
* Patients with a history of life-threatening pulmonary obstruction or a history of cystic fibrosis or bronchiectasis.
* Patients who had undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reason were to be evaluated as per exclusion criterion No. 1.
* Patients with upper respiratory tract infection in the past 6 weeks prior to the Screening visit (Visit 1, day -15) or during the run-in period.
* Patients with known hypersensitivity to anticholinergic drugs, lactose or any other components of the inhalation capsule delivery system.
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
* Patients with known narrow-angle glaucoma.
* Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count ≥ 600/mm3. A repeat eosinophil count was not to be conducted in these patients.
* Patients who were being treated with cromolyn sodium or nedocromil sodium had to stop these medications 1 month before Visit 1 (day -15).
* Patients who were being treated with antihistamines (H1 receptor antagonists) or antileukotrienes had to stop these medications 1 month before Visit 1 (day -15).
* Patients using oral corticosteroid medication at unstable doses (i.e., less than 6 weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm or Norplant®).
* Patients with history or active alcohol or drug abuse.
* Patients who had taken an investigational drug within 1 month or 10 half lives (whichever was greater) prior to Screening visit (Visit 1, day -15).
* Limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea such as arthritis in the leg, angina or claudication.
* Patients who participated in any rehabilitation program for COPD within 6 weeks prior to Visit 1 (day -15).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 1999-06; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of submaximal exercise tolerance (as measured by endurance time during a constant work rate exercise test to symptom limitation) | Day 42

SECONDARY OUTCOMES:
Endurance time after first dosing | Day 0 and 21
Determination of breathlessness (dyspnea) during constant work rate exercise test as measured by the modified Borg Scale | Day -10, -5, 0, 21 and 42
Determination of leg discomfort during constant work rate exercise test as measured by the modified Borg Scale | Day -10, -5, 0, 21 and 42
Evaluation of dynamic lung hyperinflation during exercise | Day -10, -5, 0, 21 and 42
Evaluation of dynamic hyperinflation (DH) as negative change in inspiratory capacity (IC) from rest | Day -10, -5, 0, 21 and 42
Evaluation of static lung hyperinflation | Day -10, -5, 0, 21 and 42
Evaluation of TAV (Trapped air volume) at rest | Day -10, -5, 0, 21 and 42
Evaluation of slow vital capacity (SVC) | Day -10, -5, 0, 21, 42 and 56
Evaluation of FEV1 (Forced expiratory volume in one second) | Day -10, -5, 0, 21 and 42
Evaluation of forced vital capacity (FVC) | Day -10, -5, 0, 21 and 42
Evaluation of forced expiratory flow rate between 25% and 75% of FVC which has been exhaled (FEF25-75%) | Day -10, -5, 0, 21 and 42
Evaluation of forced expiratory flow rate at 50% of FVC which has been exhaled (FEF50%) | Day -10, -5, 0, 21 and 42
Evaluation of forced expiratory flow rate at 75% of FVC which has been exhaled (FEF75%) | Day -10, -5, 0, 21 and 42
Evaluation of total lung capacity (TLC), airway resistance (Raw), and specific airway conductance (SGaw) | Day -10, -5, 0, 21 and 42
Evaluation of dyspnea using the Baseline Dyspnea Index (BDI) and Transition Dyspnoea Index (TDI) | Day 0, 21 and 42
Determination of arterial oxygen saturation (SaO2), oxygen consumption (VO2), tidal volume (VT), breathing frequency (F), and minute ventilation (VE) | Day -10, -5, 0, 21 and 42
Physicians Global Assessment | Day 0 and 42
Evaluation of COPD symptom scores | Day 0, 21 and 42
Reason for stopping constant work rate exercise | Day -15, -10, -5, 0, 21 and 42
Rescue medication use during test days | Day -15, -10, -5, 0, 21 and 42
Rescue medication use as weekly mean for number of night-time puffs (Rescni,w), daytime puffs (Rescday,w) and total daily puffs (Resctot,w) of rescue medication | until week 6